CLINICAL TRIAL: NCT03545087
Title: Pharmacokinetics of Lanabecestat (LY3314814) in Subjects With Impaired Renal Function
Brief Title: A Study of Lanabecestat in Participants With Severe Kidney Impairment Compared to Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped for futility. Phase 3 studies not likely to meet primary endpoints.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16007; I8D-MC-AZEN (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — lanabecestat; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lanabecestat Control (Experimental): Lanabecestat administered orally to participants with normal renal function
  Interventions: Drug: Lanabecestat
- Lanabecestat Severe Renal Impairment (Experimental): Lanabecestat administered orally to participants with severe renal impairment, not on dialysis
  Interventions: Drug: Lanabecestat; Drug: Iohexol

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814
Drug: Iohexol — Administered intravenously. Administration is at investigator's discretion in participants with severe renal impairment.
  Arms: Lanabecestat Severe Renal Impairment

SUMMARY:
The purpose of the study is to determine whether lanabecestat can be safely prescribed in participants with kidney impairment without a dose adjustment.

Participants will be on study for up to 6 weeks; this includes a 2-week screening and a follow-up about 10 days after final drug administration.

ELIGIBILITY:
Inclusion Criteria:

- Have a body mass index (BMI) of 19 to 40 kilograms per meter square (kg/m²)

Exclusion Criteria:

* Have a history of or current significant ophthalmic disease, particularly any eye problem involving the retina
* Have moderate or severe vitiligo or any other clinically significant disorder of skin or hair pigmentation
* Have acute unstable neuropsychiatric disease
* Have active or uncontrolled neurologic disease, or clinically significant head injury

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under The Concentration Versus Time Curve From Zero To Infinity (AUC[0-∞]) for Lanabecestat | Baseline through 168 hours after the administration of study drug
  PK: AUC(0-∞) for Lanabecestat
PK: Maximum Observed Drug Concentration (Cmax) of Lanabecestat | Baseline through 168 hours after the administration of study drug
  PK: Cmax of Lanabecestat

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Ctr., Orlando, Florida